CLINICAL TRIAL: NCT04616690
Title: Collaborative, Comparative Study on Three-dimensional Cleft Lip and Palate Morphology Prior to One-stage Cleft Repair (Warsaw/Basel)
Brief Title: Three-dimensional Cleft Lip and Palate Morphology Prior to One-stage Cleft Repair
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Institute of Mother and Child, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Benito Benitez, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: Warsaw/Basel; ch20Benitez (Other: Department of Clinical Research Basel)
Record Dates: First submitted 2020-10-25; First posted 2020-11-05 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cleft Lip and Palate; Cleft Palate; Craniofacial Deformity
Keywords: Cleft Lip and Palate; Presurgical Orthopedics; Cleft Morphology; Palatal Plate
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational cohort study of consecutive patients with cleft lip and palate deformity undergoing cleft repair at the Institute of Mother and Child in Warsaw. Cleft morphology will be captured with photo and intraoral camera before routine surgery at around 8 months. Furthermore, wound healing at 3 months postoperative will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients with orofacial cleft, who undergo routine cleft repair

Exclusion Criteria:

* missing datasets
* no signed consent for research

Ages: 6 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients eligible for this study must have an orofacial cleft which has to be treated around the age of 6-15 months.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
True Cleft Area in mm2 of Newborns With Cleft Lip and Palate at 8 Month of Age | Capture of the cleft morphology with photo and intraoral camera before routine surgery at around 8 months.
  True cleft area in mm2 will be measured at 8 month of age in newborns with cleft lip and palate.

SECONDARY OUTCOMES:
Cleft Width and Height in mm of Newborns With Cleft Lip and Palate at 8 Month of Age | Capture of the cleft morphology with photo and intraoral camera before routine surgery at around 8 months.
  Measurement of the width and height in mm of the cleft measured at 8 months of age.
Wound Healing (fistula yes or no) 3 Months After One-Stage Cleft Repair | At 3 months postoperative
  Assessment of wound healing by fistula formation at 3 months postoperative
Correlation of Cleft Width in mm and Wound Healing after One-Stage Cleft Repair | At surgery and at 3 months postoperative
  Evaluation of the correlation between cleft width in mm and wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Benito K Benitez, MD DMD, Principal Investigator — University and University Hospital of Basel; Andrzej Brudnicki, MD DDS PhD, Principal Investigator — Maxillo-facial Surgery Unit, Pediatric Surgery Clinic, Institute of Mother and Child
Locations (1):
- Institute of Mother and Child, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doray B, Badila-Timbolschi D, Schaefer E, Fattori D, Monga B, Dott B, Favre R, Kohler M, Nisand I, Viville B, Kauffmann I, Bruant-Rodier C, Grollemund B, Rinkenbach R, Astruc D, Gasser B, Lindner V, Marcellin L, Flori E, Girard-Lemaire F, Dollfus H. [Epidemiology of orofacial clefts (1995-2006) in France (Congenital Malformations of Alsace Registry)]. Arch Pediatr. 2012 Oct;19(10):1021-9. doi: 10.1016/j.arcped.2012.07.002. Epub 2012 Aug 24. French. PMID 22925539
- [Background] Wang W, Jiang B, Sun H, Ru X, Sun D, Wang L, Wang L, Jiang Y, Li Y, Wang Y, Chen Z, Wu S, Zhang Y, Wang D, Wang Y, Feigin VL; NESS-China Investigators. Prevalence, Incidence, and Mortality of Stroke in China: Results from a Nationwide Population-Based Survey of 480 687 Adults. Circulation. 2017 Feb 21;135(8):759-771. doi: 10.1161/CIRCULATIONAHA.116.025250. Epub 2017 Jan 4. PMID 28052979
- [Background] Genisca AE, Frias JL, Broussard CS, Honein MA, Lammer EJ, Moore CA, Shaw GM, Murray JC, Yang W, Rasmussen SA; National Birth Defects Prevention Study. Orofacial clefts in the National Birth Defects Prevention Study, 1997-2004. Am J Med Genet A. 2009 Jun;149A(6):1149-58. doi: 10.1002/ajmg.a.32854. PMID 19441124
- [Background] IPDTOC Working Group. Prevalence at birth of cleft lip with or without cleft palate: data from the International Perinatal Database of Typical Oral Clefts (IPDTOC). Cleft Palate Craniofac J. 2011 Jan;48(1):66-81. doi: 10.1597/09-217. Epub 2010 Apr 6. PMID 20507242
- [Background] Shaw WC, Semb G, Nelson P, Brattstrom V, Molsted K, Prahl-Andersen B, Gundlach KK. The Eurocleft project 1996-2000: overview. J Craniomaxillofac Surg. 2001 Jun;29(3):131-40; discussion 141-2. doi: 10.1054/jcms.2001.0217. PMID 11465251
- [Background] Honigmann K. One-stage closure of uni- and bilateral cleft lip and palate. Br J Oral Maxillofac Surg. 1996 Jun;34(3):214-9. doi: 10.1016/s0266-4356(96)90272-7. PMID 8818253
- [Background] Mueller AA, Zschokke I, Brand S, Hockenjos C, Zeilhofer HF, Schwenzer-Zimmerer K. One-stage cleft repair outcome at age 6- to 18-years -- a comparison to the Eurocleft study data. Br J Oral Maxillofac Surg. 2012 Dec;50(8):762-8. doi: 10.1016/j.bjoms.2012.02.002. Epub 2012 May 1. PMID 22551772
- [Background] Urbanova W, Klimova I, Brudnicki A, Polackova P, Kroupova D, Dubovska I, Rachwalski M, Fudalej PS. The Slav-cleft: A three-center study of the outcome of treatment of cleft lip and palate. Part 1: Craniofacial morphology. J Craniomaxillofac Surg. 2016 Nov;44(11):1767-1776. doi: 10.1016/j.jcms.2016.06.010. Epub 2016 Jun 17. PMID 27663676
- [Background] Brudnicki A, Piwowar W, Cudzilo D, Sawicka E. Complete unilateral cleft lip and palate operated on by means of the one-stage method - own experience. Dev Period Med. 2014;18(1):38-43. PMID 25171619
- [Background] Kozelj V. Changes produced by presurgical orthopedic treatment before cheiloplasty in cleft lip and palate patients. Cleft Palate Craniofac J. 1999 Nov;36(6):515-21. doi: 10.1597/1545-1569_1999_036_0515_cpbpot_2.3.co_2. PMID 10574670
- [Background] Kozelj V. The basis for presurgical orthopedic treatment of infants with unilateral complete cleft lip and palate. Cleft Palate Craniofac J. 2000 Jan;37(1):26-32. doi: 10.1597/1545-1569_2000_037_0026_tbfpot_2.3.co_2. PMID 10670886
- [Background] Nalabothu P, Benitez BK, Dalstra M, Verna C, Mueller AA. Three-Dimensional Morphological Changes of the True Cleft under Passive Presurgical Orthopaedics in Unilateral Cleft Lip and Palate: A Retrospective Cohort Study. J Clin Med. 2020 Mar 31;9(4):962. doi: 10.3390/jcm9040962. PMID 32244361